CLINICAL TRIAL: NCT00557245
Title: Parallel Comparison of Tenofovir and Emtricitabine/Tenofovir Pre-Exposure Prophylaxis to Prevent HIV-1 Acquisition Within HIV-1 Discordant Couples
Brief Title: Pre-Exposure Prophylaxis to Prevent HIV-1 Acquisition Within HIV-1 Discordant Couples
Acronym: Partners PrEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Connie Celum, Professor, School of Medicine, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00000172; IND 75,365;; 07-7454-A-01
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: HIV-1 Infections; HIV Infections
Keywords: HIV infection; HIV uninfected partners; Double Blind; Placebo; Seroconversion; TDF; FTC TDF; Safety; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; HIV Seropositivity | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tenofovir Disoproxil Fumarate (TDF) (Active Comparator): TDF 300 mg tablet, once daily + Placebo FTC/TDF orally, once daily.
  Interventions: Drug: Tenofovir Disoproxil Fumarate (TDF)
- Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) (Active Comparator): FTC/TDF - 200 mg tablet, once daily + Placebo TDF orally, once daily
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF)
- Placebo (Placebo Comparator): Placebo TDF + Placebo FTC/TDF orally, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate (TDF) — TDF 300 mg tablet, once daily + Placebo FTC/TDF orally, once daily.
  Other Names: Viread + Placebo Truvada
  Arms: Tenofovir Disoproxil Fumarate (TDF)
Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) — FTC/TDF - 200 mg tablet, once daily + Placebo TDF orally, once daily
  Other Names: Truvada + Placebo Viread
  Arms: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF)
Drug: Placebo — Placebo TDF & Placebo FTC/TDF, 1 tablet each daily.
  Other Names: Placebo + Placebo
  Arms: Placebo

SUMMARY:
Randomized, blinded, placebo-controlled trial to demonstrate if pre-exposure prophylaxis decreases HIV-1 acquisition among HIV-1 uninfected individuals within HIV-1 discordant couples.

DETAILED DESCRIPTION:
HIV-1 uninfected individuals within HIV-1 discordant partnerships are at high-risk for HIV-acquisition. The majority of HIV-1 transmissions to adults in Africa occur within stable, HIV-1 discordant couples.

Pre-exposure chemoprophylaxis, in which an HIV-1 uninfected individual at high risk for contracting HIV-1 takes antiretroviral medications to maintain blood and genital drug levels sufficient to prevent HIV-1 acquisition, has been proposed as a potential HIV-1 prevention strategy.

This study was a randomized, blinded, placebo-controlled trial to demonstrate if pre-exposure prophylaxis decreases HIV-1 acquisition among HIV-1 uninfected individuals within HIV-1 discordant couples. The HIV-1 uninfected partner was randomized in a 1:1:1 ratio to one of three arms: once daily Tenofovir Disoproxil Fumarate (TDF), Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) or Placebo.

Couples were followed up to 36 months; the HIV uninfected partner attended monthly visits and the HIV infected partner quarterly visits. All participants received a comprehensive package of HIV prevention services including individual and couples counseling, free condoms, and male circumcision referrals.

Participants who seroconverted during follow-up stopped the study drug but continued with follow-up.

ELIGIBILITY:
Inclusion Criteria for HIV-1 uninfected partner:

* Partner within an HIV-1 discordant heterosexual relationship
* One partner meets study eligibility for HIV-1 uninfected study participant and the other partner meets study eligibility criteria for HIV-1 infected participant
* Plan to remain in the relationship for the duration of the study period
* Adequate renal, hepatic & hematologic function
* Negative Hepatitis B surface antigen test
* Willing and able to provide written informed consent & locator information

Exclusion Criteria for HIV-1 uninfected partner:

* Current pregnancy, or planning to become pregnant during the study period
* Currently breastfeeding
* Concurrent enrollment in another HIV-1 vaccine or prevention trial
* Receiving ongoing antiretroviral therapy
* Repeated positive urine dipstick tests for glycosuria or proteinuria
* Active and serious infections
* History of pathological bone fractures not related to trauma

Inclusion Criteria for HIV-1 infected partner:

* Partner within an HIV-1 discordant heterosexual relationship
* One partner meets study eligibility for HIV-1 uninfected study participant and the other partner meets study eligibility criteria for HIV-1 infected participant
* HIV-1 infected based on positive EIA
* No history of any clinical AIDS-defining diagnoses
* Plan to remain in the relationship for the duration of the study period
* Willing and able to provide written informed consent & locator information

Exclusion Criteria for HIV-1 infected partner:

* Current use of antiretroviral therapy
* Concurrent enrollment in another HIV-1 treatment trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4758 (Actual)
Dates: Start 2008-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum,, MD, MPH, Study Chair — University of Washington; Jared Baeten, MD, PhD, Study Director — University of Washington
Locations (9):
- Kenya (4):
  - Moi University - Indiana University, Eldoret
  - CMR, Kemri-UCSF, Kisumu
  - Kenyatta National Hospital/University of Nairobi, Nairobi
  - Partners in Prevention - Thika, Thika
- Uganda (5):
  - Kabwohe Clinical Research Center, Bushenyi
  - Infectious Diseases Institute, Jinja
  - Partners House-Infectious Disease Institute Ltd, Kampala
  - The AIDS Support Organization (TASO), Mbale
  - The AIDS Support Organization - Tororo Field Station, Tororo

REFERENCES:
- [Background] Mujugira A, Baeten JM, Donnell D, Ndase P, Mugo NR, Barnes L, Campbell JD, Wangisi J, Tappero JW, Bukusi E, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kidoguchi L, Panteleeff D, Krows M, Shah H, Revall J, Morrison S, Ondrejcek L, Ingram C, Coombs RW, Lingappa JR, Celum C; Partners PrEP Study Team. Characteristics of HIV-1 serodiscordant couples enrolled in a clinical trial of antiretroviral pre-exposure prophylaxis for HIV-1 prevention. PLoS One. 2011;6(10):e25828. doi: 10.1371/journal.pone.0025828. Epub 2011 Oct 5. PMID 21998703
- [Result] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Derived] Saha A, Escuduero J, Layouni T, Richardson B, Hou S, Mugo N, Mujugira A, Celum C, Baeten JM, Lingappa J, John-Stewart GC, LaCourse SM, Shah JA. Mycobacterium tuberculosis-Specific T-Cell Responses Are Impaired During Late Pregnancy With Elevated Biomarkers of Tuberculosis Risk Postpartum. J Infect Dis. 2022 May 4;225(9):1663-1674. doi: 10.1093/infdis/jiab614. PMID 34929030
- [Derived] Mugo NR, Eckert L, Magaret AS, Cheng A, Mwaniki L, Ngure K, Celum C, Baeten JM, Galloway DA, Wamalwa D, Wald A. Quadrivalent HPV vaccine in HIV-1-infected early adolescent girls and boys in Kenya: Month 7 and 12 post vaccine immunogenicity and correlation with immune status. Vaccine. 2018 Nov 12;36(46):7025-7032. doi: 10.1016/j.vaccine.2018.09.059. Epub 2018 Oct 5. PMID 30297124
- [Derived] Mackelprang RD, Bamshad MJ, Chong JX, Hou X, Buckingham KJ, Shively K, deBruyn G, Mugo NR, Mullins JI, McElrath MJ, Baeten JM, Celum C, Emond MJ, Lingappa JR; Partners in Prevention HSV/HIV Transmission Study and the Partners PrEP Study Teams. Whole genome sequencing of extreme phenotypes identifies variants in CD101 and UBE2V1 associated with increased risk of sexually acquired HIV-1. PLoS Pathog. 2017 Nov 6;13(11):e1006703. doi: 10.1371/journal.ppat.1006703. eCollection 2017 Nov. PMID 29108000
- [Derived] Mugwanya K, Baeten J, Celum C, Donnell D, Nickolas T, Mugo N, Branch A, Tappero J, Kiarie J, Ronald A, Yin M, Wyatt C; Partners PrEP Study Team. Low Risk of Proximal Tubular Dysfunction Associated With Emtricitabine-Tenofovir Disoproxil Fumarate Preexposure Prophylaxis in Men and Women. J Infect Dis. 2016 Oct 1;214(7):1050-7. doi: 10.1093/infdis/jiw125. Epub 2016 Mar 29. PMID 27029778
- [Derived] Mugwanya KK, Wyatt C, Celum C, Donnell D, Mugo NR, Tappero J, Kiarie J, Ronald A, Baeten JM; Partners PrEP Study Team. Changes in glomerular kidney function among HIV-1-uninfected men and women receiving emtricitabine-tenofovir disoproxil fumarate preexposure prophylaxis: a randomized clinical trial. JAMA Intern Med. 2015 Feb;175(2):246-54. doi: 10.1001/jamainternmed.2014.6786. PMID 25531343
- [Derived] Baeten JM, Donnell D, Mugo NR, Ndase P, Thomas KK, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kidoguchi L, Coombs RW, Hendrix C, Marzinke MA, Frenkel L, Haberer JE, Bangsberg D, Celum C; Partners PrEP Study Team. Single-agent tenofovir versus combination emtricitabine plus tenofovir for pre-exposure prophylaxis for HIV-1 acquisition: an update of data from a randomised, double-blind, phase 3 trial. Lancet Infect Dis. 2014 Nov;14(11):1055-1064. doi: 10.1016/S1473-3099(14)70937-5. Epub 2014 Oct 7. PMID 25300863
- [Derived] Mugo NR, Hong T, Celum C, Donnell D, Bukusi EA, John-Stewart G, Wangisi J, Were E, Heffron R, Matthews LT, Morrison S, Ngure K, Baeten JM; Partners PrEP Study Team. Pregnancy incidence and outcomes among women receiving preexposure prophylaxis for HIV prevention: a randomized clinical trial. JAMA. 2014 Jul 23-30;312(4):362-71. doi: 10.1001/jama.2014.8735. PMID 25038355
- [Derived] Celum C, Morrow RA, Donnell D, Hong T, Hendrix CW, Thomas KK, Fife KH, Nakku-Joloba E, Mujugira A, Baeten JM; Partners PrEP Study Team. Daily oral tenofovir and emtricitabine-tenofovir preexposure prophylaxis reduces herpes simplex virus type 2 acquisition among heterosexual HIV-1-uninfected men and women: a subgroup analysis of a randomized trial. Ann Intern Med. 2014 Jul 1;161(1):11-9. doi: 10.7326/M13-2471. PMID 24979446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Started | 1589 | 1583 | 1586
Completed | 1577 | 1571 | 1574
Not Completed | 12 | 12 | 12
Not completed — Lost to Follow-up | 7 | 8 | 10
Not completed — Ineligible | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants, less those who were found to be ineligible (n=11)
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo | Total
Number analyzed (Participants) | 1584 | 1579 | 1584 | 4747
Age, Customized [Number; unit: participants]
  18-24 years | 184 | 177 | 172 | 533
  25-34 years | 721 | 690 | 688 | 2099
  35-44 years | 480 | 498 | 513 | 1491
  45 years and older | 199 | 214 | 211 | 624
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 598 | 566 | 621 | 1785
  Male | 986 | 1013 | 963 | 2962
Region of Enrollment [Number; unit: participants]
  Kenya | 700 | 698 | 697 | 2095
  Uganda | 884 | 881 | 887 | 2652
Percentage of participants who had unprotected sex in the past month [Number; unit: percentage of participants] — The percentage of participants who had any unprotected sex acts in the prior month.
  percentage of participants | 27.9 | 26.3 | 25.8 | 26.7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of HIV-1 Seroconversion Among HIV-1 Uninfected Participants
Description: The efficacy of once daily PrEP in preventing HIV-1 acquisition among uninfected heterosexuals in HIV-1 discordant partnerships, measured by calculating the HIV incidence per 100 person-years in each of three arms.
Time Frame: Up to 36 months
Population: All randomized participants, less those who were found to ineligible (n=11), less those found to be infected at enrollment (n=14), and less those who did not return for any follow-up (n=25).
Measure: Number (95% Confidence Interval); unit: events per 100 person years
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 1572 | 1568 | 1568
events per 100 person years | 0.65 [0.38 to 1.05] | 0.50 [0.27 to 0.85] | 1.99 [1.49 to 2.62]
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; We used Cox regression stratified according to site, to estimate the relative rates of time to first positive HIV-1 serologic test; Test type: Superiority or Other; p < 0.001, Regression, Cox — The a priori threshold was 0.05; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.19 to 0.56] — Placebo arm is the reference group
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Cox — The a priori threshold was 0.05; Hazard Ratio (HR) = 0.25, 95% CI 2-sided [0.13 to 0.45] — Placebo arm is the reference group

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Safety of daily TDF or FTC/TDF among HIV-1 uninfected individuals randomized to TDF or FTC/TDF compared to those randomized to placebo measured as the number of participants with Serious Adverse Events (SAEs) during follow-up.
Time Frame: Up to 36 months
Population: Randomized participants, less those found to be ineligible (n=11)
Measure: Number; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 1584 | 1579 | 1584
Participants | 118 | 115 | 118
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; Test type: Superiority or Other; p = 0.89, Fisher Exact

3. Secondary Outcome: Study Drug Adherence: Total Number of Study Drug Doses Taken of the Total Dispensed Doses.
Description: Adherence to study medication as assessed by pill count at follow-up visits. We assessed the total number of doses taken of the total dispensed doses.
Time Frame: Up to 36 months
Measure: Number; unit: percentage of doses taken of dispensed
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 1571 | 1565 | 1570
percentage of doses taken of dispensed | 97 | 97 | 97

4. Secondary Outcome: Study Drug Adherence: Self-reported Missed Doses of Study Drug
Description: Adherence to study drug measured as the percentage of visits when participants reported missing 1) any dose of study drug in the prior month and 2) 2 or more consecutive doses of study drug.
Time Frame: Up to 36 months
Population: Participants with self-reported adherence.
Measure: Number; unit: percentage of visits
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 1549 | 1552 | 1551
percentage of visits
  Missed any doses | 15 | 15 | 15
  Missed 2+ consecutive doses | 4 | 4 | 4

5. Secondary Outcome: Number of Seroconverters With an HIV-1 Mutation Conferring Resistance to TDF or FTC
Description: HIV-1 resistance as measured by the number of seroconverters who had an HIV-1 reverse transcriptase mutation (K65R, K70E, M184I, or M184V) conferring resistance to TDF or FTC. These mutation types were pre-defined. Plasma samples for resistance testing were collected at the visit seroconversion was first detected and again at a visit within 1 month of seroconversion. Mutations detected at either of those visits are reported.
  Both seroconverters found to have a resistance mutation had been HIV infected at enrollment (TDF arm: n=1; FTC-TDF arm: n=1).
Time Frame: Up to 36 months
Population: Participants who seroconverted during the Partners PrEP trial, including those who were retrospectively found to be HIV infected at enrollment (TDF arm: n=5; FTC-TDF arm: n=3; placebo arm: n=6). For 4 of 96 HIV-1 seroconverters (TDF arm: n=2; FTC-TDF arm: n=1; placebo arm: n=1) HIV-1 RNA was unable to be amplified for HIV-1 resistance testing.
Measure: Number; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 20 | 15 | 57
Participants | 1 | 1 | 0

6. Secondary Outcome: Number of Participants With a Sexually Transmitted Infection (STI) During Follow-up
Description: Prevalence of STIs measured as the number of participants with a positive test result for N. gonorrhoeae, C. trachomatis, or T. vaginalis during follow-up. Participants were tested for STIs at annual follow-up visits and at intervening visits at which the participant presented with symptoms of an STI. Assessment for symptomatic sexually transmitted infections was conducted quarterly.
  N. gonorrhoeae and C. trachomatis testing were by APTIMA Combo 2 (Gen-Probe) or COBAS Amplicor (Roche Diagnostics). T. vaginalis testing was by APTIMA TV TMA (Gen-Probe) or In Pouch TV (Biomed Diagnostics).
Time Frame: Up to 36 months
Population: Randomized participants, less those found to be ineligible (n=11)
Measure: Number; unit: participants
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 1584 | 1579 | 1584
participants | 102 | 76 | 85
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; Test type: Superiority or Other; p = 0.24, Regression, Logistic; Generalized estimating equations, with logistic link and robust standard errors to adjust for individual correlation over time
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; Test type: Superiority or Other; p = 0.49, Regression, Logistic; [statistical method as in outcome 6, analysis 1]

7. Secondary Outcome: Prevalence of Unprotected Sex During Follow-up
Description: Sexual risk behavior of participants, measured as the percentage of visits when participants reported having unprotected sex during follow-up.
Time Frame: Up to 36 months
Population: All randomized participants, less those found to be ineligible (n=11).
Measure: Number; unit: percentage of visits
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 1584 | 1579 | 1584
percentage of visits | 14 | 13 | 13
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; Test type: Superiority or Other; p = 0.32, Regression, Logistic; Generalized estimating equations, logistic link, with robust standard errors
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; Test type: Superiority or Other; p = 0.66, Regression, Logistic; Generalized estimating equations, logistic link, with robust standard errors

8. Secondary Outcome: Congenital Abnormalities Among Infants Born to Female Participants Taking Study Drug.
Description: Infant outcomes measured as the number of live-born infants born to female participants taking study drug that had any congenital anomalies.
Time Frame: Up to 36 months
Population: Randomized female participants, less those found to be ineligible (n=7)
Measure: Number; unit: Number of live-born infants
Units Other Than Participants: live-born infants
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 595 | 565 | 621
Number analyzed (live-born infants) | 81 | 47 | 66
Number of live-born infants | 4 | 4 | 5
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; Test type: Superiority or Other; p = 0.51, Regression, Logistic; Generalized estimating equations with logistic link to account for multiple pregnancies and multiple births
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; Test type: Superiority or Other; p = 0.86, Regression, Logistic; generalized estimating equations with logistic link to account for multiple pregnancies and multiple births

9. Secondary Outcome: Length Among Infants Born to Female Participants Taking Study Drug
Description: The slope of the linear model of the growth of infants (length) during the entirety of follow-up. The length of the infant was measured as a z-score, in terms of standard deviations from the age and gender specific median using the World Health Organization growth curve, accounting for skewness. The slope, representing the change over time of the z-score, was calculated using all available z-scores over 12 months and regressing against study month.
Time Frame: up to 12 months
Population: Infants born to women taking study drug during follow-up
Measure: Number; unit: z-score difference per study month
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 81 | 47 | 66
z-score difference per study month | -0.006 | 0.036 | -0.033
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; Test type: Superiority or Other; p = 0.42, Mixed Models Analysis; linear mixed-effects model
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis; Linear mixed-effects model; Slope Difference over time = 0.07 — Placebo arm is the reference group

10. Secondary Outcome: Weight Among Infants Born to Female Participants Taking Study Drug
Description: The slope of the linear model of the growth of infants (weight) during the entirety of follow-up. The weight of the infant was measured as a z-score, in terms of standard deviations from the age and gender specific median using the World Health Organization growth curve, accounting for skewness. The slope, representing the change over time of the z-score, was calculated using all available z-scores over 12 months and regressing against study month.
Time Frame: up to 12 months
Population: Infants born to women taking study drug during follow-up
Measure: Number; unit: z-score difference per study month
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 81 | 47 | 66
z-score difference per study month | -0.021 | 0.009 | -0.056
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Linear mixed effects model
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Linear mixed effects model

11. Secondary Outcome: Head Circumference Among Infants Born to Female Participants Taking Study Drug
Description: The slope of the linear model of the growth of infants (head circumference) during the entirety of follow-up. The head circumference of the infant was measured as a z-score, in terms of standard deviations from the age and gender specific median using the World Health Organization growth curve, accounting for skewness. The slope, representing the change over time of the z-score, was calculated using all available z-scores over 12 months and regressing against study month.
Time Frame: up to 12 months
Population: Infants born to women taking study drug during follow-up
Measure: Number; unit: z-score difference per study month
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Number analyzed (Participants) | 81 | 47 | 66
z-score difference per study month | -0.057 | -0.005 | -0.079
Statistical Analysis 1: Comparison: Tenofovir Disoproxil Fumarate (TDF) vs Placebo; Test type: Superiority or Other; p = 0.35, Mixed Models Analysis; Linear mixed effects model
Statistical Analysis 2: Comparison: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs Placebo; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Linear mixed effects model

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | Tenofovir Disoproxil Fumarate (TDF) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | Placebo
Serious Adverse Events (participants affected / at risk) | 118/1584 | 115/1579 | 118/1584
Other Adverse Events (participants affected / at risk) | 1306/1584 | 1316/1579 | 1297/1584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tenofovir Disoproxil Fumarate (TDF) (N=1584) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) (N=1579) | Placebo (N=1584)
ANKYLOGLOSSIA CONGENITAL (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0)
EXOMPHALOS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
HYPOSPADIAS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
POLYDACTYLY (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
SYNDACTYLY (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
BLINDNESS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
OPTIC NEUROPATHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
ACUTE ABDOMEN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
PEPTIC ULCER (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (4)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
TOOTH DEVELOPMENT DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOLVULUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 2 (2) | 0 (0)
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE HIV INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ANAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
APPENDICITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
BREAST ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRUCELLOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL MALARIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CERVICITIS (Infections and infestations) | 1/598 (1) | 0/566 (0) | 0/621 (0)
DYSENTERY (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
FEBRILE INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
GASTROENTERITIS SHIGELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HORDEOLUM (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MALARIA (Infections and infestations) | 28 (31) | 28 (30) | 37 (40)
ORCHITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
PELVIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 3/598 (3) | 0/566 (0) | 0/621 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SALPINGITIS (Infections and infestations) | 0/598 (0) | 0/566 (0) | 1/621 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TYPHOID FEVER (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
CATARACT TRAUMATIC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CHEMICAL EYE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
DRUG TOXICITY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ELECTROCUTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 3 (3)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INDUCED ABORTION HAEMORRHAGE (Injury, poisoning and procedural complications) | 0/598 (0) | 0/566 (0) | 1/621 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 6 (6)
SCIATIC NERVE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 3 (3)
STRUCK BY LIGHTNING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 2 (2) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 2 (2) | 2 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 5 (5) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 13 (15) | 18 (20) | 10 (10)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 5 (5) | 4 (5)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
FRACTURE MALUNION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/598 (0) | 0/566 (0) | 1/621 (1)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/598 (0) | 1/566 (1) | 0/621 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 7/598 (7) | 8/566 (8) | 6/621 (6)
ANTEPARTUM HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 0/598 (0) | 1/566 (1) | 0/621 (0)
NORMAL DELIVERY (Pregnancy, puerperium and perinatal conditions) | 5/598 (5) | 2/566 (2) | 2/621 (2)
PERINEAL LACERATION (Pregnancy, puerperium and perinatal conditions) | 1/598 (1) | 0/566 (0) | 0/621 (0)
POSTPARTUM HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 0/598 (0) | 0/566 (0) | 1/621 (1)
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 1/598 (1) | 0/566 (0) | 1/621 (1)
PROLONGED LABOUR (Pregnancy, puerperium and perinatal conditions) | 0/598 (0) | 1/566 (1) | 0/621 (0)
ACUTE PSYCHOSIS (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SCHIZOPHRENIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1/986 (1) | 1/1013 (1) | 0/963 (0)
CERVIX DISORDER (Reproductive system and breast disorders) | 1/598 (1) | 0/566 (0) | 0/621 (0)
FALLOPIAN TUBE CYST (Reproductive system and breast disorders) | 0/598 (0) | 0/566 (0) | 1/621 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 1/598 (1) | 0/566 (0) | 0/621 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0/598 (0) | 1/566 (1) | 1/621 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SCAR PAIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
VICTIM OF CRIME (Social circumstances) | 1 (1) | 0 (0) | 1 (1)
COLOSTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tenofovir Disoproxil Fumarate (TDF) (N=1584) | Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) (N=1579) | Placebo (N=1584)
NEUTROPHIL COUNT DECREASED (Investigations) | 598 (1109) | 686 (1322) | 577 (1076)
BLOOD PHOSPHORUS DECREASED (Investigations) | 440 (763) | 460 (785) | 473 (787)
MALARIA (Infections and infestations) | 290 (371) | 267 (356) | 280 (352)
HAEMOGLOBIN DECREASED (Investigations) | 259 (384) | 230 (335) | 231 (331)
PLATELET COUNT DECREASED (Investigations) | 190 (306) | 188 (305) | 177 (298)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 125 (147) | 159 (189) | 142 (169)
BLOOD BICARBONATE DECREASED (Investigations) | 123 (142) | 118 (130) | 135 (148)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 108 (117) | 91 (107) | 114 (133)
URINARY TRACT INFECTION (Infections and infestations) | 105 (121) | 86 (96) | 103 (122)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 93 (138) | 103 (146) | 96 (124)
BLOOD CREATININE INCREASED (Investigations) | 76 (99) | 107 (126) | 86 (108)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 90 (103) | 87 (104) | 73 (85)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 50 (59) | 71 (93) | 64 (83)
BLOOD BILIRUBIN INCREASED (Investigations) | 56 (82) | 49 (64) | 63 (88)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 59/598 (71) | 48/566 (55) | 55/621 (62)
DIARRHOEA (Gastrointestinal disorders) | 48 (56) | 37 (39) | 39 (41)
PROTEINURIA (Renal and urinary disorders) | 40 (47) | 36 (46) | 34 (43)
GASTROENTERITIS (Infections and infestations) | 33 (36) | 32 (34) | 30 (32)
GENITAL ULCERATION (Reproductive system and breast disorders) | 26 (29) | 35 (48) | 34 (38)
TYPHOID FEVER (Infections and infestations) | 32 (39) | 28 (31) | 23 (24)
SYPHILIS (Infections and infestations) | 28 (30) | 27 (31) | 23 (24)
GASTRITIS (Gastrointestinal disorders) | 20 (22) | 28 (31) | 24 (28)
ABDOMINAL PAIN (Gastrointestinal disorders) | 23 (23) | 22 (23) | 24 (24)
CELLULITIS (Infections and infestations) | 26 (27) | 12 (13) | 26 (27)
HYPERTENSION (Vascular disorders) | 19 (20) | 14 (18) | 30 (42)
URETHRITIS (Infections and infestations) | 26 (33) | 16 (16) | 20 (22)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 19 (19) | 27 (28)
URETHRAL DISCHARGE (Renal and urinary disorders) | 17 (20) | 21 (23) | 18 (22)
PNEUMONIA (Infections and infestations) | 16 (17) | 17 (19) | 21 (23)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 18 (18) | 19 (19) | 16 (17)
COUGH (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 20 (21) | 11 (12)
PHARYNGITIS (Infections and infestations) | 16 (16) | 18 (18) | 15 (15)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 13/598 (14) | 19/566 (20) | 17/621 (17)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 17 (17) | 16 (16) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes